CLINICAL TRIAL: NCT03452696
Title: Clinical Trial to Evaluate the Gastric Tolerability and Efficacy of the Food Supplement of Microencapsulated Calcium Carbonate vs Conventional Calcium Carbonate and Calcium Citrate
Brief Title: Clinical Trial to Evaluate the Tolerability and Efficacy of Microencapsulated Calcium Carbonate
Acronym: CALCIMIP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Palacios (Other)
Collaborators: Nexentia S.A.S. (Unknown)
Responsible Party: Principal Investigator, Dr. Santiago Palacios, Principal Investigator, Instituto Palacios
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CALCIMIP18
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Hypocalcemia; Dietary
MeSH Terms: conditions — Hypocalcemia

STUDY DESIGN:
Who Masked: Participant
Masking Description: Women
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Calcium supplement 10/90 (Experimental): Microencapsulated calcium, 1389 mg orally (10% protein and 90% calcium carbonate, corresponding to 500 mg of calcium element per tablet). There will be 2 doses of 1389 mg each orally, to make a total contribution of 1,000 mg. of calcium element.
  Interventions: Dietary Supplement: Calcium supplement
- Calcium supplement 5/95 (Experimental): Microencapsulated calcium1316 mg orally (5% protein and 95% calcium carbonate, corresponding to 500 mg of calcium element per tablet). There will be 2 shots of 1,316 mg each orally, to make a total contribution of 1,000 mg. calcium element
  Interventions: Dietary Supplement: Calcium supplement
- Calcium carbonate supplement (Active Comparator): 1,250 mg orally (500 mg of calcium element). There will be 2 doses of 1,250 mg. each orally, to make a total contribution of 1,000 mg. of calcium element.
  Interventions: Dietary Supplement: Calcium supplement
- Calcium citrate supplement (Active Comparator): 1,500 mg orally (315 mg of calcium element). There will be 2 taken orally, to make a total contribution of 945 mg. calcium element
  Interventions: Dietary Supplement: Calcium supplement

INTERVENTIONS:
Dietary Supplement: Calcium supplement — Calcium supplement for low contribution of elemental calcium in the daily diet

SUMMARY:
Interventional Clinical trial with food supplement, randomized, double-blind, comparative between microencapsulated calcium, calcium carbonate salts standardized and calcium citrate, in a population of postmenopausal women, lasting 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal woman
* Low contribution of elemental calcium in the daily diet

Exclusion Criteria:

* Hypersensitivity to the active substances or to any of the excipients
* Renal insufficiency
* History of kidney or urinary stones
* Use in the last month of diuretics (furosemide, ethacrynic acid), aluminum salts and / or thyroid hormones
* Use of any other drug or experimental device during the 30 days prior to the selection

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women
Enrollment: 208 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
Gastric symptoms | 1 month
  Using the Gastrointestinal Symptom Rating Scale (GRS). The scale measures constipation, diarrhea, windiness, swelling, nausea, reflux, pain and burning. The patient will have to choose the most appropriate response among those proposed. "Not at all" is the better outcome and "very strong discomfort" is the worst outcome

SECONDARY OUTCOMES:
Changes in bone markers | Basal and 1 month
  Bone Marker Analysis (CTx and P1NP) will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Palacios, PI, Principal Investigator — Instituto Palacios
Locations (1):
- Instituto Palacios, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided